CLINICAL TRIAL: NCT04814303
Title: Adductor Canal Block Versus Periarticular Infiltration Effect on Functional Outcome In Patients Undergoing Total Knee Replacement
Brief Title: Impact of Adductor Canal Block on Functional Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abbas Hassan, lectrure of Anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Adductor canal block in TKR
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ITM (Active Comparator): spinal anesthesia will be induced with heavy bupivacaine 0.5% 12.5-15 mg (2.5-3 mL) at L3-4 or L4-5 inter-vertebral and Intrathecal morphine 150 μg will be added.
  Interventions: Procedure: Intrathecal morphine
- ACB (Active Comparator): spinal anesthesia will be induced with heavy bupivacaine 0.5% 12.5-15 mg (2.5-3 mL) at L3-4 or L4-5 inter-vertebral and Intrathecal morphine 150 μg will be added. The block will be performed in the mid adductor canal to block both the saphenous and the nerve to vastus medialis. After skin infiltration with 1 to 2 mL of 2% lidocaine, an 80-mm, 22-gauge, the short-bevel echogenic needle is advanced in-plane with the ultrasound beam in an anterior-to-posterior direction until the tip is located within the adductor canal deep to the vastoadductor membrane. After negative aspiration, 1-2 mL of local anesthetic is injected to confirm the proper injection plane. The study solution will be injected within the canal adjacent to the femoral artery. Patients in this group received 30 mL of 0.25% bupivacaine with 1:400,000 epinephrine and 4 mg dexamethasone.
  Interventions: Procedure: Intrathecal morphine; Procedure: Adductor Canal block
- PAI (Active Comparator): spinal anesthesia will be induced with heavy bupivacaine 0.5% 12.5-15 mg (2.5-3 mL) at L3-4 or L4-5 inter-vertebral and Intrathecal morphine 150 μg will be added. PAI intra-operatively will be performed with 150 mL of 0.25% bupivacaine with 1:400,000 epinephrine, 30 mg of ketorolac, and 8 mg dexamethasone.
  Interventions: Procedure: Intrathecal morphine; Procedure: Peri-articular Infilteration

INTERVENTIONS:
Procedure: Intrathecal morphine — After applying standard monitoring of pulse oximetry, ECG, NIBP; while the patient in the sitting position following complete sterile aseptic condition after sterilization bovine bethidine spinal anesthesia will be induced with heavy bupivacaine 0.5% 12.5-15 mg (2.5-3 mL) at L3-4 or L4-5 inter-vertebral levels using a 25- gauge Whitacre needle. Intrathecal morphine 150 μg will be added to patients of both groups. Supplemental oxygen will be administered via a simple face mask.
Procedure: Adductor Canal block — The block will be performed in the mid adductor canal to block both the saphenous and the nerve to vastus medialis. After skin infiltration with 1 to 2 mL of 2% lidocaine, an 80-mm, 22-gauge, short-bevel echogenic needle is advanced in plane with the ultrasound beam in an anterior-to-posterior direction until the tip is located within the adductor canal deep to the vastoadductor membrane. After negative aspiration, 1-2 mL of local anesthetic is injected to confirm the proper injection plane. The study solution will be injected within the canal adjacent to the femoral artery. Patients in group 1 received 30 mL of 0.25% bupivacaine with 1:400,000 epinephrine and 4 mg dexamethasone.
  Arms: ACB
Procedure: Peri-articular Infilteration — the surgeon will perform the PAI intra-operatively; 150 mL of 0.25% bupivacaine with 1:400,000 epinephrine, 30 mg of ketorolac, and 8 mg dexamethasone. Half of the solution will be administered into the posterior capsule and posterior soft tissues of the knee under direct vision after osteotomy but before insertion of the implants. The remaining half of the solution will be administered into the anterior soft tissues after placement of the implants and before skin closure. All local infiltration will be carried out while a thigh tourniquet (used to limit surgical bleeding) was inflated at a pressure of 300 to 350 mm Hg.
  Arms: PAI

SUMMARY:
TKA involves extensive bone resection as well as soft tissue excision and therefore is associated with profound postoperative pain. Adequate analgesia after TKA is therefore considered paramount to facilitate early hospital discharge and effective functional recovery.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee has become a major public health issue and imposes a significant healthcare burden and accounts for high annual hospitalizations. Chronic OA of the knee may lead to reduced physical fitness, mobility disability with a resultant increased risk of cardio-metabolic comorbidity and early mortality. Total knee arthroplasty (TKA) is indicated in severe cases to improve long-term pain and function. (1) TKA involves extensive bone resection as well as soft tissue excision and therefore is associated with profound postoperative pain. (2) Inadequate perioperative pain control may prolong hospitalization, hinder early rehabilitation, and is also a strong predictor of persistent pain beyond 3 months. (3) Adequate analgesia after TKA is therefore considered paramount to facilitate early hospital discharge and effective functional recovery. (4) The recently introduced adductor canal block (ACB) typically covers the anterio-medial aspect of the knee and preserves quadriceps function, which presumably enhances postoperative rehabilitation by allowing patients to actively participate in knee movement. The relative effectiveness of this ACB technique added to intrathecal morphine is limited to a single study (1) in which assessment of short-term functional recovery was done and dexamethasone was neither included in the LIA solution nor perineurally in the ACB. Thus, we hypothesize that adductor canal block as an adjunct to intrathecal morphine will have a better impact on functional recovery than peri-articular infiltration.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist class ( ASA) I - III
* BMI 18-35 kg/m2
* Scheduled for primary unilateral TKR

Exclusion Criteria:

* Known allergy to local anesthetics
* Contraindication to adductor canal block e.g. infection at the site of injection
* Contraindication to spinal anesthesia e.g. coagulopathy.
* Patients with pre-existing motor or sensory deficits in lower extremities.
* Patients who are morbidly obese (BMI≥35) because ultrasound-guided regional anesthesia could be technically difficult.
* Bilateral or revision total knee replacement
* Insulin or noninsulin-dependent diabetes mellitus.
* systemic corticosteroid use within 30-days of surgery

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
"Timed Up and Go" test (TUG) | 48 hours
  reflects the time it takes a subject to stand up from a standard-height armchair, walk 3 m, walk back to the chair, and sit down.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) at rest | 72 hours
  will be used to assess knee pain intensity
Visual analogue scale (VAS) at movement | 72 hours
  will be used to assess knee pain intensity
Time to first analgesic request | 72 hours
  the first time the patient ask for analgesia
Total analgesic consumption | 72 hours
  Total consumption of postoperative rescue analgesics (total of paracetamol doses) will be recorded